CLINICAL TRIAL: NCT00695708
Title: Training-induced Cerebral Reorganization in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Rockstroh Brigitte, Prof. Dr., University of Konstanz
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: RO 805/14
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2008-06

CONDITIONS: Schizophrenia
Keywords: schizophrenia; neuroplasticity; sensory gating; cognitive impairment; MEG; Disorders with Psychotic Features
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BFT (Experimental): 20 schizophrenic patients
  Interventions: Behavioral: Brain Fitness Program
- CP (Active Comparator): 19 schizophrenic patients
  Interventions: Behavioral: Cogpack
- HCG (No Intervention): 20 healthy age and sex matched subjects

INTERVENTIONS:
Behavioral: Brain Fitness Program — Computer-aided cognitive program designed for intensive training of auditory perception, memory and attention
  Arms: BFT
Behavioral: Cogpack — Computer-aided cognitive program for cognitive abilities
  Arms: CP

SUMMARY:
The purpose of this study is to reveal the effects of computer-aided cognitive-auditory training on cerebral reorganization in schizophrenia.

DETAILED DESCRIPTION:
Impairment in cognitive functions is one of the main symptoms in schizophrenia and is currently one of the challenges in the treatment of the disease.

In this study we compare effects of two computer-aided training programs. One focused on auditory perception and processing as a basic ability underlying higher order information processing.

The other training involves a variability of cognitive abilities.

Both trainings are computer-aided and time-intensive, including up to twenty sessions within four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia and disorders with psychotic features
* Intact hearing abilities

Exclusion Criteria:

* Mental retardation
* Age over 60
* Insufficient German language knowledge

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Event related potential MEG, test scores in word fluency and verbal learning tasks | pre and post intervention

SECONDARY OUTCOMES:
Symptom severity, GAF score | pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Rockstroh, Prof. Dr., Study Chair — University of Konstanz, Department of Psychology
Locations (1):
- University of Konstanz, Konstanz, Baden Württenberg, Germany

REFERENCES:
- [Derived] Popov T, Jordanov T, Rockstroh B, Elbert T, Merzenich MM, Miller GA. Specific cognitive training normalizes auditory sensory gating in schizophrenia: a randomized trial. Biol Psychiatry. 2011 Mar 1;69(5):465-71. doi: 10.1016/j.biopsych.2010.09.028. Epub 2010 Nov 18. PMID 21092939